CLINICAL TRIAL: NCT07399184
Title: Comparison of the Effects of Ibuprofen on Cerebral Oxygenation, Postoperative Cognitive Dysfunction, and Delirium in One-Lung Ventilation
Brief Title: Effect of Perioperative IV Ibuprofen on Cerebral Oxygenation and Postoperative Cognition During One-Lung Ventilation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Elif Bengi SENER, Professor of Anesthesiology, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IBU2025
Record Dates: First submitted 2026-02-02; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Delirium; Cerebral Oxygen Saturation; Postoperative Cognitive Dysfunction (POCD)
Keywords: cerebral oxygenation; near infrared spectroscopy; thoracic anesthesia; postoperative delirium; one lung ventilation; ibuprofen
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications | interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: This study is conducted using a parallel-group interventional study model. Eligible participants are randomly assigned in a 1:1 ratio to one of two groups: the ibuprofen intervention group or the control group. Randomization is performed using a computer-generated allocation sequence and implemented via sequentially numbered, opaque, sealed envelopes to ensure allocation concealment.
  The intervention is applied perioperatively, and participants remain in their assigned group throughout the study with no crossover between groups. Outcomes are assessed and compared between groups in parallel over the defined intraoperative and postoperative follow-up period. The study is designed as prospective, single-center, randomized, controlled, and single-blind, consistent with a parallel assignment model.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBUPROFEN (GROUP B) (Experimental): In the study, patients will be randomized into two groups (Group B: ibuprofen group; Group C: control group). Patients in Group B will receive 400 mg intravenous ibuprofen administered by the anesthesia research resident 15 minutes before the surgical incision. Group B patients will also receive postoperative intravenous ibuprofen at a dose of 400 mg three times daily. No intraoperative or postoperative ibuprofen treatment will be administered to patients in Group C.
  Interventions: Drug: ibuprofen
- CONTROL (GROUP C) (No Intervention): In this study, patients will be randomized into two groups (Group B: ibuprofen group; Group C: control group). Patients in Group B will receive 400 mg IV ibuprofen administered by the anesthesia research resident 15 minutes before the surgical incision. Group B patients will also receive postoperative IV ibuprofen at a dose of 400 mg three times daily. No intraoperative or postoperative ibuprofen treatment will be administered to patients in Group C.

INTERVENTIONS:
Drug: ibuprofen — In the study, patients in Group B will receive a single intraoperative dose of 400 mg IV ibuprofen, followed by postoperative administration of 400 mg IV ibuprofen three times daily for 24 hours. We hypothesize that, by benefiting from the anti-inflammatory effects of ibuprofen, intraoperative cerebral oxygenation will be preserved, thereby reducing the incidence of postoperative delirium and cognitive dysfunction.
  Other Names: IV ibuprofen
  Arms: IBUPROFEN (GROUP B)

SUMMARY:
This study compares the effects of ibuprofen administered during surgery and within the first 24 hours after surgery, versus no ibuprofen, on cerebral oxygenation, postoperative changes in consciousness (postoperative delirium and cognitive dysfunction), length of stay in the intensive care unit, and the incidence of postoperative pain, nausea, vomiting, and pruritus in patients undergoing lung lobectomy or segmentectomy using a closed (video-assisted) method (VATS - video-assisted thoracoscopic surgery), in whom one-lung ventilation is applied.

The aim of this study is to evaluate the effects of ibuprofen on cerebral oxygenation, postoperative cognitive changes, and delirium in patients undergoing one-lung ventilation.

DETAILED DESCRIPTION:
During one-lung ventilation (OLV) in thoracic surgery, cerebral oxygenation may decrease due to hypoxia, and this condition can be evaluated noninvasively using near-infrared spectroscopy (NIRS) . The ability of near-infrared light to penetrate tissues and be absorbed by oxyhemoglobin and deoxyhemoglobin forms the basic principle of measuring regional cerebral oxygen saturation. With this method, the balance between oxygen supply and demand in cerebral tissue can be continuously and dynamically assessed in real time. During measurements, it is assumed that the blood volume within the venous, capillary, and arterial compartments of the brain remains constant. Therefore, cerebral oximeters provide an average value reflecting oxygenation across these compartments. Low regional cerebral oxygen saturation values have been associated with cerebral hypoxia and/or ischemia.

Cerebral hypoxia is a well-known risk factor for postoperative delirium (POD) . While anesthesia has traditionally been considered the primary cause of postoperative delirium, animal studies suggest that surgery-induced inflammation may be an important contributor to neurological disorders associated with postoperative delirium. The peripheral inflammatory response affects the brain and contributes to the pathogenesis of postoperative delirium. Cytokines, particularly IL-1β, TNF-α, and IL-6, are believed to interact with the brain . The mechanisms by which peripheral cytokines reach the brain are thought to involve the blood-brain barrier or the circumventricular regions. These peripheral cytokines trigger microglia-derived cytokine synthesis, leading to a cycle of neuroinflammation. A recent meta-analysis of human observational studies has shown that both peripheral and cerebrospinal fluid (CSF) inflammatory markers, such as CRP and IL-6, are associated with postoperative delirium and postoperative cognitive dysfunction . Postoperative delirium occurs at a rate of 10-20% and prolongs hospital stay by 2-3 days and intensive care unit stay by approximately 2 days .

Due to surgery-induced systemic inflammatory responses, patients may also experience postoperative cognitive dysfunction (POCD). POCD is usually observed in the immediate postoperative period and manifests as a transient cognitive impairment. This condition may range from fatigue, social withdrawal, and decreased concentration to severe cognitive dysfunction. POCD may also lead to fluctuating levels of consciousness and disturbances in the sleep-wake cycle.

The incidence of POCD is highest among elderly patients. It has been observed in up to 40% of patients aged 60 years and older who undergo surgery. Although postoperative cognitive fluctuations are often not considered alarming, POCD is thought to predict the future onset of dementia and may contribute to chronic neurodegeneration with repeated surgical procedures.

Increases in pro-inflammatory cytokines during surgery trigger short-term cognitive impairment. Additionally, evidence from animal studies suggests that TNF-α-mediated dysfunction of the blood-brain barrier and migration of leukocytes into the hippocampus may lead to memory impairment. Nonsteroidal anti-inflammatory drugs (NSAIDs) are widely used as a component of multimodal postoperative analgesia, and it has been suggested that these agents may prevent postoperative delirium by directly alleviating neuroinflammation. The primary mechanism of action of NSAIDs is the inhibition of the cyclooxygenase (COX) enzyme responsible for prostaglandin synthesis. The constitutive isoform, COX-1, plays a role in intercellular signaling and tissue homeostasis, whereas COX-2, which is induced in inflammatory cells, is responsible for the production of prostanoids involved in inflammation. Ibuprofen exerts its effects by inhibiting both COX-1 and COX-2. Inhibition of COX-1 may be responsible for undesirable gastrointestinal side effects ; however, inhibition of COX-2 provides ibuprofen with its analgesic, antipyretic, and anti-inflammatory properties. In a study conducted by Huang et al. in mice, perioperative use of ibuprofen was shown to improve cognitive performance, reduce systemic inflammation, and decrease glial activation . In clinical settings, preoperative administration of intravenous ibuprofen has been shown to improve postoperative cognitive function in association with reduced levels of cytokines, cortisol, and catecholamines. Additionally, another study demonstrated that the use of the NSAID flurbiprofen increased PaO₂ levels .

However, no studies have investigated the effects of ibuprofen on PaO₂, cerebral oxygenation, postoperative delirium, or postoperative cognitive dysfunction in patients undergoing one-lung ventilation.The aim of this study is to investigate the effects of administered intravenous ibuprofen on intraoperative cerebral oxygenation and subsequent postoperative cognitive function changes in patients undergoing lobectomy or segmentectomy via VATS with one-lung ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years
* American Society of Anesthesiologists (ASA) Physical Status Classification System I-III
* Patients scheduled for lobectomy or segmentectomy via Video-Assisted Thoracic Surgery (VATS ) with one-lung ventilation
* New York Heart Association (NYHA) class I-II
* Patients who have been informed about the study and have provided written informed consent will be included.

Exclusion Criteria:

* Patients younger than 18 years or older than 75 years
* History of alcohol or substance abuse
* Patients with chronic NSAID use and/or NSAID use within the last 30 days, or NSAID allergy
* Allergy to other drugs used in the study (e.g., bupivacaine)
* ASA Physical Status IV-V
* Severe hearing, visual, or speech impairment
* Dementia, Alzheimer's disease, or psychiatric disorders (psychosis, bipolar disorder, schizophrenia)
* History of previous head trauma
* Chronic liver disease
* Pregnancy
* History of cerebrovascular disease
* Moderate-to-severe chronic obstructive pulmonary disease (COPD) (predicted FEV₁ <50%)
* GFR <60 mL/min/1.73 m²
* Patients who do not provide written informed consent
* Conditions that may cause inaccurate cerebral oximetry readings (subdural and/or extracranial hematoma, intracranial arteriovenous shunts, hyperbilirubinemia)
* Patients undergoing emergency surgery
* Patients in whom surgery is initiated as thoracotomy or converted to thoracotomy
* Patients unable to complete the preoperative MMSE (total score ≤24) will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Right and left intraoperative cerebral oxygenation values (rScO₂) | preoperative and intraoperative
  The primary outcome of this study is the preoperative and intraoperative right and left regional cerebral oxygenation values. Cerebral oxygenation is measured using near-infrared spectroscopy (NIRS). The ability of near-infrared light to penetrate biological tissues and to be absorbed by oxyhemoglobin and deoxyhemoglobin constitutes the basic principle of regional cerebral oxygen saturation measurement. Using this method, the balance between oxygen supply and demand in cerebral tissue can be continuously evaluated in real time. During measurements, it is assumed that the blood volume within the venous, capillary, and arterial compartments of the brain remains constant. Therefore, cerebral oximeters provide an average value reflecting the oxygenation of these compartments. Low regional cerebral oxygen saturation values have been associated with cerebral hypoxia and/or ischemia.

SECONDARY OUTCOMES:
Postoperative cognitive dysfunction (MMSE score) | until the end of postoperative day 2 and preoperative day
  Cognitive functions in the preoperative and postoperative periods will be assessed using the Mini-Mental State Examination (MMSE) for patients with at least 5 years of education, and the MMSE for uneducated individuals for those with less than 5 years of education. Patients unable to complete the test (total score ≤24) will be excluded from the study.
Postoperative delirium score (NU-DESC) | until the end of postoperative day 2
  NU-DESC is a delirium screening tool. A total score of 2 or higher will be considered clinically significant for delirium.
Postoperative Resting and activity NRS score (Numeric Rating Scale) | until the end of postoperative day 1
  Patients' pain will be assessed using the Resting and activity NRS (Numeric Rating Scale), scored from 0 to 10. Rescue analgesia will be administered if the score is 4 or higher.
Postoperative nausea and vomiting status | until the end of postoperative day 1
  Nausea and vomiting will be assessed using the Verbal Descriptive Scale (VDS), with scores ranging from 0 to 4. Accordingly, patients with a score of 3 or higher will receive IV ondansetron at a dose of 0.05 mg/kg.

CONTACTS AND LOCATIONS:
Overall Officials: Canan ASAR SAHIN, Study Director — Ondokuz Mayıs University Faculty of Medicine Department of Anesthesiology and Reanimation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen L, Chen JQ, Yang XL, Hu JC, Gao W, Chai XQ, Wang D. Corrigendum: Flurbiprofen used in one-lung ventilation improves intraoperative regional cerebral oxygen saturation and reduces the incidence of postoperative delirium. Front Psychiatry. 2023 Jun 6;14:1228369. doi: 10.3389/fpsyt.2023.1228369. eCollection 2023. PMID 37346900
- [Background] Tang L, Kazan R, Taddei R, Zaouter C, Cyr S, Hemmerling TM. Reduced cerebral oxygen saturation during thoracic surgery predicts early postoperative cognitive dysfunction. Br J Anaesth. 2012 Apr;108(4):623-9. doi: 10.1093/bja/aer501. Epub 2012 Feb 5. PMID 22311364
- [Background] Hayashi K, Yamada Y, Ishihara T, Tanabe K, Iida H. Comparison of regional cerebral oxygen saturation during one-lung ventilation under desflurane or propofol anesthesia: A randomized trial. Medicine (Baltimore). 2022 Oct 14;101(41):e30030. doi: 10.1097/MD.0000000000030030. PMID 36254073
- [Background] Liu Z, Jin Y, Wang L, Huang Z. The Effect of Ciprofol on Postoperative Delirium in Elderly Patients Undergoing Thoracoscopic Surgery for Lung Cancer: A Prospective, Randomized, Controlled Trial. Drug Des Devel Ther. 2024 Feb 5;18:325-339. doi: 10.2147/DDDT.S441950. eCollection 2024. PMID 38344256